CLINICAL TRIAL: NCT04616950
Title: Impact of the COVID-19 Epidemic on the Hospital Journey of Patients With Cancer of the Digestive System: Description of Typical Pathways and Simulation Model
Brief Title: Impact of the COVID-19 Epidemic on the Hospital Journey of Patients With Cancer of the Digestive System
Acronym: KOVID
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: KOVID
Record Dates: First submitted 2020-11-04; First posted 2020-11-05 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Covid19; Cancer
MeSH Terms: conditions — COVID-19; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The hospital care of patients with cancerous pathology is part of a multidisciplinary care path that includes many stages. The treatment conditions in this course vary depending on the reasons that led to suspect the existence of a cancerous pathology: accidental discovery, screening, warning signs (sometimes expressed in an acute form) or referral for treatment in charge after the diagnosis has already been made. As soon as the patient presents to the hospital, various expertises are mobilized to establish the diagnosis, carry out the extension assessment and assess the comorbidities and conditions that may have an impact on the choice of treatments. During this initial evaluation, each file is evaluated in a Multidisciplinary Consultation Meeting to define the optimal therapeutic strategy which will often include several stages involving surgery, radiotherapy, medical oncology (chemotherapy, immunotherapy, targeted therapy, etc. hormone therapy), interventional radiology, and / or supportive oncological care (nutrition, pain treatment, correction of metabolic abnormalities, palliative care, etc.). This treatment path is considered to be very complex and the fluidity of its organization determines the processing times.

The management of patients in a cancer department may vary depending on the organization specific to each hospital. The health crisis induced by the COVID-19 epidemic, associated with the containment measures put in place from March 19 to May 11, 2020, have limited the use of patients in hospitals, even for emergency activities. It has also led to a reorganization of scheduled activities within establishments, with a concentration of resources around unscheduled care, in particular COVID patients. In many establishments, the other activities were, for many, deprogrammed with postponed appointments. The impact of this epidemic on the hospital journey of patients with cancerous pathology is the subject of questions at the national level. The delays in diagnosis and treatment induced have possibly had an impact on the quality of the care and on the delays with, as a corollary, a possible loss of opportunity for the patient.

DETAILED DESCRIPTION:
The hospital care of patients with cancerous pathology is part of a multidisciplinary care path that includes many stages. The treatment conditions in this course vary depending on the reasons that led to suspect the existence of a cancerous pathology: accidental discovery, screening, warning signs (sometimes expressed in an acute form) or referral for treatment in charge after the diagnosis has already been made. As soon as the patient presents to the hospital, various expertises are mobilized to establish the diagnosis, carry out the extension assessment and assess the comorbidities and conditions that may have an impact on the choice of treatments. During this initial evaluation, each file is evaluated in a Multidisciplinary Consultation Meeting to define the optimal therapeutic strategy which will often include several stages involving surgery, radiotherapy, medical oncology (chemotherapy, immunotherapy, targeted therapy, etc. hormone therapy), interventional radiology, and / or supportive oncological care (nutrition, pain treatment, correction of metabolic abnormalities, palliative care, etc.). This treatment path is considered to be very complex and the fluidity of its organization determines the processing times.

The management of patients in a cancer department may vary depending on the organization specific to each hospital. Most often, this is secondary management after the patient has been taken care of by the emergency department - the diagnosis is then suspected but not yet established - or tertiary by a medical specialty service or surgical - the diagnosis is then established and part of the treatment, in particular surgical, has already been carried out. Primary care by addressing from correspondents outside the hospital directly to medical oncology is possible but rarer, particularly at Saint-Joseph Hospital. The first treatment by the oncology service is therefore carried out after a fairly complex preliminary hospital course, the duration of which is likely to vary depending on the number and complexity of each of the preliminary stages. The duration of the different stages of the care pathway is a very important element in the quality of the care because unjustified delays can impact on the therapeutic results.

The health crisis induced by the COVID-19 epidemic, associated with the containment measures put in place from March 19 to May 11, 2020, have limited the use of patients in hospitals, even for emergency activities. It has also led to a reorganization of scheduled activities within establishments, with a concentration of resources around unscheduled care, in particular COVID patients. In many establishments, the other activities were, for many, deprogrammed with postponed appointments. The impact of this epidemic on the hospital journey of patients with cancerous pathology is the subject of questions at the national level. The delays in diagnosis and treatment induced have possibly had an impact on the quality of the care and on the delays with, as a corollary, a possible loss of opportunity for the patient.

Within the Paris Saint-Joseph Hospital Group, which strongly participated in the management of the pandemic over the period from March 15 to June 15, 2020, observations were made compared to the same period in 2019:

* An 80% drop in day hospital stays for gastrology and proctology endoscopy
* A 60% drop in stays in digestive and proctological surgery (full hospitalization, week or day)
* A 40% decrease in emergency room consultations, as well as an activity focused on the care of COVID patients
* A decrease in consulting activities
* A reorganization of the healthcare offer: block restricted to emergencies, limitation of endoscopy activity and imaging activity.

During this epidemic period, a specific organization was adopted within the oncology department which made it possible to immediately continue the chemotherapy protocols initiated. Among the measures put in place, the investigators can cite the compulsory wearing of a mask and hand washing with hydro-alcoholic solution for patients and caregivers, the restriction of accompanying persons and visits with protection conditions, the sanctuarization of the service without PCR patients COVID + or symptomatically suspected, individual monitoring of each suspected or COVID + patient, follow-up teleconsultations, etc. These measures put in place from March 19, 2020 have made it possible to maintain the treatments as defined in the SPC for patients already admitted to the service. However, the hospital journey of patients upstream of their medical oncology treatment has been severely impacted by the COVID-19 epidemic. In this context, the objectification of the disturbances induced by the epidemic is of interest from an epidemiological and public health point of view. It is also likely to nourish reflection on securing the organization of this course within the establishment. Our work falls within this perspective. The investigators were more particularly interested in the impact of the COVID-19 epidemic on the care pathway of digestive cancer patients whose treatment path is complex before arriving in the oncology department for their first treatment therapeutic load.

A first phase of the study will consist of the description of the hospital journey of patients with cancer of the digestive system requiring management by the medical oncology department of the Paris Saint-Joseph hospital. Two periods will be considered (before / after COVID) in order to assess the impact of the COVID-19 epidemic on the routes studied.

A second phase of the study will consist of modeling the hospital journey based on observations made during the period preceding the COVID-19 epidemic. This modeling will make it possible to simulate the impact of any "disruptions" that would be exerted on one or other of the components of the course (less patient use in the hospital, limited access to various expertise and technical facilities). The objective pursued in the long term would be to have a tool that would allow this impact to be anticipated and to test in silico the potential effectiveness of the measures that could be implemented to limit its extent.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years
* Patients with primary cancer of the digestive system: cancer of the esophagus, stomach, small intestine, colon, rectosigmoid junction, rectum, anal canal, liver , gall bladder, bile ducts and pancreas;
* Patients hospitalized for the first time in the medical oncology department in full hospitalization, week or day;
* Patients hospitalized between January 1, 2019 and October 31, 2020
* French-speaking patient

Exclusion Criteria:

* Patients with secondary cancer or a relapse of cancer of the digestive system
* Patients who do not require hospitalization in medical oncology
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under legal protection
* Patient objecting to the use of their medical data in the context of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary cancer of the digestive system: cancer of the esophagus, stomach, small intestine, colon, rectosigmoid junction, rectum, anal canal, liver , gall bladder, bile ducts and pancreas; were hospitalized for the first time in the oncology department within the Paris Saint Joseph Hospital Group, between January 1, 2019 and October 31, 2020.
Sampling Method: Non-Probability Sample
Enrollment: 274 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
Hospital course of patients with cancer of the digestive system | Day 1
  This outcome corresponds to the basis of the delay, measured as a continuous quantitative variable, in number of days between entry into the course and the first inpatient treatment in the medical oncology department.

SECONDARY OUTCOMES:
Modeling of the hospital journey based on observations made during the period preceding the COVID-19 epidemic | Day 1
  This outcome corresponds to the characterization of the course will be studied: entry points, expertise mobilized, arrangement of the different "components" of the course and the time between each of them.

CONTACTS AND LOCATIONS:
Overall Officials: Anne BURONFOSSE, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, Groupe Hospitalier Paris Saint-Joseph, France

REFERENCES:
- [Result] Belle A, Barret M, Bernardini D, Tarrerias AL, Bories E, Costil V, Denis B, Gincul R, Karsenti D, Koch S, Laquiere A, Lecomte T, Quentin V, Rahmi G, Robaszkiewicz M, Vaillant E, Vanbiervliet G, Vienne A, Dumeiran F, Gronier O, Chaussade S; French Society of Digestive Endoscopy (Societe Francaise d'Endoscopie Digestive). Impact of the COVID-19 pandemic on gastrointestinal endoscopy activity in France. Endoscopy. 2020 Dec;52(12):1111-1115. doi: 10.1055/a-1201-9618. Epub 2020 Jul 8. PMID 32557489
- [Result] Soreide K, Hallet J, Matthews JB, Schnitzbauer AA, Line PD, Lai PBS, Otero J, Callegaro D, Warner SG, Baxter NN, Teh CSC, Ng-Kamstra J, Meara JG, Hagander L, Lorenzon L. Immediate and long-term impact of the COVID-19 pandemic on delivery of surgical services. Br J Surg. 2020 Sep;107(10):1250-1261. doi: 10.1002/bjs.11670. Epub 2020 Apr 30. PMID 32350857
- [Result] Grosclaude P, Azria D, Guimbaud R, Thibault S, Daubisse-Marliac L, Cartron G, Renaudie MJ, Dalbies PA, Delord JP, Bauvin E. [COVID-19 impact on the cancer care structuration: Example of the multidisciplinary team meeting dedicated to oncology in Occitanie]. Bull Cancer. 2020 Jul-Aug;107(7-8):730-737. doi: 10.1016/j.bulcan.2020.05.001. Epub 2020 May 18. French. PMID 32425210
- [Result] Sud A, Jones ME, Broggio J, Loveday C, Torr B, Garrett A, Nicol DL, Jhanji S, Boyce SA, Gronthoud F, Ward P, Handy JM, Yousaf N, Larkin J, Suh YE, Scott S, Pharoah PDP, Swanton C, Abbosh C, Williams M, Lyratzopoulos G, Houlston R, Turnbull C. Collateral damage: the impact on outcomes from cancer surgery of the COVID-19 pandemic. Ann Oncol. 2020 Aug;31(8):1065-1074. doi: 10.1016/j.annonc.2020.05.009. Epub 2020 May 19. PMID 32442581
- [Result] Gelman A, Rubin DB. Markov chain Monte Carlo methods in biostatistics. Stat Methods Med Res. 1996 Dec;5(4):339-55. doi: 10.1177/096228029600500402. PMID 9004377